CLINICAL TRIAL: NCT01502150
Title: Data Collection of Normal Tissue Toxicity for Proton Therapy for Pediatrics
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PCR05-0208
Record Dates: First submitted 2011-12-21; First posted 2011-12-30 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Pediatric Cancer
Keywords: Pediatric Cancer; Proton Radiation Therapy; Proton beam radiotherapy; PBT; Data Collection; Database; Acute and late normal tissue toxicities; Dosimetric data; Toxicity data
MeSH Terms: conditions — Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Proton Therapy Patients: Data collection of MDACC patients under the age of 18 treated with proton radiotherapy. Proton dosimetry data collection, corresponding radiation dose distribution and imaging data in order to correlate normal tissue response with dose distribution.
  Interventions: Other: Data Collection; Other: Dose Distribution Data Collection

INTERVENTIONS:
Other: Data Collection — Information collected from follow-up visits post proton radiation therapy yearly or more often, and test results for at least 10-15 years.
Other: Dose Distribution Data Collection — Data collection of complete plan information, including dose distribution, beam configuration and images, computed tomography (CT) images acquired on multiple days and 4D CT's for respiratory correlated imaging.

SUMMARY:
The goal of this research study is to collect information on the side effects of proton therapy and the details of proton treatment plans so that researchers can develop a method to predict the risk of side effects and to improve the planning and delivery of proton treatment for patients in the future.

DETAILED DESCRIPTION:
If you agree to take part in this study, researchers will gather information about your treatment and treatment outcomes and store it electronically in a database. By carefully evaluating the data about your treatment, researchers may improve proton treatment for patients in the future. There will be no change to your recommended standard of care and follow-up studies. The treatment information and follow-up information will be stored in a database. The information will then be available at a later date for researchers to study. The database will be stored on a secure information network, and only those people who are involved with this research and who have prior approval from the study doctor will have access to it.

Researchers will request information from the follow-up visits that you have as part of your standard of care yearly or more often and test results for at least 10-15 years. The tests may be performed at other clinics, but MD Anderson researchers will request that the results be sent to them at MD Anderson.

This is an investigational study. Proton radiotherapy is FDA approved. Researchers hope to enroll all children who will be treated with proton radiotherapy at MD Anderson on this study so that as much information as possible will be gathered. Up to 1000 patients will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria

1. All patients under the age of 18 who are treated with PBT will be eligible to participate in this trial.
2. Signed informed consent must be obtained from the patient or patient's representative prior to study enrollment.

Exclusion Criteria:

1. Pregnant females are not eligible.
2. Patient or patient's parent or legal guardian representative is unable or unwilling to give informed consent.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric cancer patients receiving proton radiation therapy at MD Anderson Cancer Center in Houston, Texas
Sampling Method: Non-Probability Sample
Enrollment: 798 (Actual)
Dates: Start 2005-06-16 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Data Collection From Pediatric Patients Undergoing Proton Radiation Therapy | 15 years
  For each acute normal-tissue endpoint considered, analyses will be performed using the maximum toxicity score per patient within the 90-day follow-up. For each late normal-tissue endpoint considered, analyses will be performed using censored time-to-event data corresponding to specified levels of injury (e.g. time to a specific grade >= 2 late toxicity).

CONTACTS AND LOCATIONS:
Overall Officials: Arnold dela Cruz Paulino, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org